CLINICAL TRIAL: NCT06351163
Title: Minimally Invasive Surgical Management for Pediatric Intussusception: A Retrospective Cohort Study on the Long-Term Outcome
Brief Title: Minimally Invasive Surgical Management for Pediatric Intussusception: A Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: National Children's Hospital, Vietnam (Other)
Collaborators: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Principal Investigator, Nguyen Thanh Quang, Pediatric Surgeon, National Children's Hospital, Vietnam
Other Study IDs: 1451_03/BVNTW-VNCSKTE
Record Dates: First submitted 2024-04-01; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Intussusception
Keywords: Intussusception; Minimally-invasive; Laparoscopic; Children; Pediatric; Air enema; Pneumatic reduction
MeSH Terms: conditions — Intussusception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intussusception: Pediatric patients exhibiting clinical signs and symptoms of intussusception between January 2016 and December 2020 that fit in with the inclusion criteria of the study.
  Interventions: Procedure: Laparoscopic reduction; Procedure: Transumbilical mini-open reduction

INTERVENTIONS:
Procedure: Laparoscopic reduction — A 1cm longitudinal transumbilical incision was made to insert a 5mm trocar for laparoscope placement. CO2 was injected at 10mmHg and a flow rate of 3L. Two 5-mm working trocars were inserted in the lower right and left abdomen under direct visualization, along with two grasping forceps. The ascending colon was manipulated to locate the intussusception mass. Atraumatic graspers were alternately utilized on the ascending colon to mobilize the intussusceptum, pushing it downward towards the cecum. The first visible part of the terminal ileum was grasped and pulled outward and downward, along with its mesentery, using the right grasper, while the left grasper pulled the intussusceptum's neck in the opposite direction. If resistance was encountered, the terminal ileum could be held with the left hand while the right grasper widened the intussusceptum's neck. After reduction, the intestines were examined for necrosis and possible lead points, followed by routine appendectomy and ileopexy.
Procedure: Transumbilical mini-open reduction — If laparoscopic reduction alone was unsuccessful or if bowel resection was required, the intussusceptum was fixed with grasping forceps and brought to the umbilicus for MOR. A 2cm transumbilical incision was created, and a skin retractor was inserted. The underlying fascia was longitudinally extended upward and downward along the linea alba. Upon division of the peritoneum, the actual opening could be expanded up to 5cm, while maintaining the skin incision at 2cm. If the initial incision site proved insufficient for exploration, lateral division of the rectus muscle around the umbilicus on both sides could be performed without cutting the skin, thereby enlarging the surgical field. Manual reduction of the intussusceptum was subsequently carried out, along with bowel resection and anastomosis as indicated.

SUMMARY:
Intussusception is the primary cause of intestinal obstruction in children aged 3 months to 5 years, leading to significant morbidity and mortality rates. Most cases involve the ileocolic region and can often be resolved through air enema, with a success rate of up to 95%. Surgical intervention becomes necessary if pneumatic reduction fails or is not recommended. Traditionally, manual reduction required a large incision on the right side of the abdomen. However, the advancement of minimally invasive techniques, such as the laparoscopic approach (LAP), has become increasingly popular for managing intussusception. LAP offers benefits such as reduced surgical trauma and shorter operative times compared to open procedures. Nevertheless, the adoption of LAP remains controversial due to challenges like limited working space in children and variability in the affected bowel segment. This study aims to investigate the safety and feasibility of LAP and mini-open reduction (MOR) techniques in treating idiopathic intussusception in pediatric patients.

DETAILED DESCRIPTION:
Intussusception, the leading cause of intestinal obstruction in children aged 3 months to 5 years, significantly impacts morbidity and mortality rates. Most cases involve the ileocolic region and are typically amenable to resolution via air enema, achieving success rates of up to 95%. Surgical intervention becomes necessary in cases where pneumatic reduction fails or is contraindicated. Historically, the manual reduction required a substantial right-sided transverse incision. However, the advancement of minimally invasive approaches in pediatric surgery, particularly the laparoscopic approach (LAP), has gained traction in managing intussusception. LAP offers the advantages of decreased surgical trauma and shorter operative durations compared to open procedures. Nevertheless, the adoption of laparoscopic intervention for intussusception remains contentious due to challenges such as limited operative space in pediatric patients and variability in the affected bowel segment, impeding widespread acceptance. This study aims to investigate the safety and feasibility of laparoscopic (LAP) and mini-open reduction (MOR) techniques in managing idiopathic intussusception in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with idiopathic intussusception, admitted to the National Children's Hospital between January 2016 and December 2020, exhibiting clinical signs and symptoms consistent with intussusception, and confirmed by ultrasound.
* Fluoroscopy-guided pneumatic reduction was performed, allowing a maximum of three attempts.
* Patients unresponsive to pneumatic reduction underwent laparoscopic reduction (LAP).
* If LAP failed to manage the intussusceptum, conversion to transumbilical mini-open reduction (MOR) was initiated.
* Patients deemed unsuitable for air enema reduction due to a grossly distended abdomen or compromised cardiopulmonary function, making them unlikely to tolerate pneumoperitoneum, were also directed towards MOR.
* Patients with a history of previous intussusception episodes requiring reduction.
* Patients displaying clinical instability with signs of peritonitis or intestinal perforation requiring conventional laparotomy.
* Patients presenting with pathologic lead points.
* Patients who had complications, such as perforation, during pneumatic reduction.

Exclusion Criteria:

* Patients in critical condition or suspected of bowel perforation and peritonitis
* Patients who did not meet the criteria for air enema reduction due to significant abdominal distension or compromised cardiopulmonary function

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: From January 2016 to December 2020, a group of pediatric patients displaying clinical manifestations suggestive of intussusception, coupled with positive ultrasound results, were admitted to the emergency department of the Vietnam National Children's Hospital. The patients underwent pneumatic reduction up to three attempts, with LAP being indicated if air enema reduction failed.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2024-03 (Actual)

PRIMARY OUTCOMES:
Operating time | through study completion (5 years)
  The average operating time (minutes) recorded between the two operating techniques (MOR or LAP)
Intraoperative complications | through study completion (5 years)
  Instances of complications occurred during both operating techniques (MOR or LAP)
Immediate postoperative complications | through study completion (5 years)
  Instances of complication occurred immediately subsequent to the operation utilizing either MOR or LAP
Time to feed | through study completion (5 years)
  The average amount of time (days) for the patient to tolerate feeding post-operation (MOR or LAP)
Hospital stays | through study completion (5 years)
  The average amount of time (days) for the patient to get discharged post-operation (MOR or LAP)
Recurrence rate | through study completion (5 years)
  Instances when signs or symptoms of intussusception re-occurred after receiving treatment via operation (MOR or LAP)
Long-term complication rate | through study completion (5 years)
  Instances of complications occurred post-operation found on subsequent follow-ups for patients treated with either MOR or LAP

CONTACTS AND LOCATIONS:
Overall Officials: Quang T Nguyen, Principal Investigator — Department of Pediatric Surgery, The National Hospital of Pediatrics, Hanoi, Vietnam
Locations (2):
- Vietnam (2):
  - The National Hospital of Pediatrics, Hanoi
  - Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang PC, Duh YC, Fu YW, Hsu YJ, Wei CH. Single-incision laparoscopic surgery for idiopathic intussusception in children: Comparison with conventional laparoscopy. J Pediatr Surg. 2019 Aug;54(8):1604-1608. doi: 10.1016/j.jpedsurg.2018.07.010. Epub 2018 Jul 21. PMID 30121127
- [Background] Bailey KA, Wales PW, Gerstle JT. Laparoscopic versus open reduction of intussusception in children: a single-institution comparative experience. J Pediatr Surg. 2007 May;42(5):845-8. doi: 10.1016/j.jpedsurg.2006.12.037. PMID 17502196
- [Background] Attoun MA, Albalawi SMD, Ayoub A, Alnasser AK, Alkaram EH, Khubrani FA, Alzahrani KJ, Alatawi KA, Almutairi N, Alnami AG. The Management of Intussusception: A Systematic Review. Cureus. 2023 Nov 27;15(11):e49481. doi: 10.7759/cureus.49481. eCollection 2023 Nov. PMID 38152810
- [Background] Cuckow PM, Slater RD, Najmaldin AS. Intussusception treated laparoscopically after failed air enema reduction. Surg Endosc. 1996 Jun;10(6):671-2. doi: 10.1007/BF00188527. PMID 8662412
- [Background] Kelley-Quon LI, Arthur LG, Williams RF, Goldin AB, St Peter SD, Beres AL, Hu YY, Renaud EJ, Ricca R, Slidell MB, Taylor A, Smith CA, Miniati D, Sola JE, Valusek P, Berman L, Raval MV, Gosain A, Dellinger MB, Somme S, Downard CD, McAteer JP, Kawaguchi A. Management of intussusception in children: A systematic review. J Pediatr Surg. 2021 Mar;56(3):587-596. doi: 10.1016/j.jpedsurg.2020.09.055. Epub 2020 Oct 6. PMID 33158508
- [Background] Wu P, Huang P, Fu Y, Lv Y, Feng S, Lou Y. Laparoscopic versus Open Reduction of Intussusception in Infants and Children: A Systematic Review and Meta-analysis. Eur J Pediatr Surg. 2022 Dec;32(6):469-476. doi: 10.1055/s-0042-1749437. Epub 2022 Jun 10. PMID 35688449
- [Background] Delgado-Miguel C, Garcia A, Delgado B, Munoz-Serrano A, Miguel-Ferrero M, Camps JI, Lopez-Santamaria M, Martinez L. Incidental appendectomy in surgical treatment of ileocolic intussusception in children. Is it safe to perform? Cir Pediatr. 2022 Oct 1;35(4):165-171. doi: 10.54847/cp.2022.04.16. English, Spanish. PMID 36217786
- [Background] Liu T, Wu Y, Xu W, Liu J, Sheng Q, Lv Z. A retrospective study about incidental appendectomy during the laparoscopic treatment of intussusception. Front Pediatr. 2022 Sep 6;10:966839. doi: 10.3389/fped.2022.966839. eCollection 2022. PMID 36147812
- [Background] Zhang Y, Wang Y, Zhang Y, Hu X, Li B, Ming G. Laparoscopic Ileopexy Versus Laparoscopic Simple Reduction in Children with Multiple Recurrences of Ileocolic Intussusception: A Single-Institution Retrospective Cohort Study. J Laparoendosc Adv Surg Tech A. 2020 May;30(5):576-580. doi: 10.1089/lap.2019.0641. Epub 2020 Apr 2. PMID 32240037
- [Background] Loukas M, Pellerin M, Kimball Z, de la Garza-Jordan J, Tubbs RS, Jordan R. Intussusception: an anatomical perspective with review of the literature. Clin Anat. 2011 Jul;24(5):552-61. doi: 10.1002/ca.21099. Epub 2011 Jan 25. PMID 21268121
- [Background] Li B, Sun CX, Chen WB, Zhang FN. Laparoscopic Ileocolic Pexy as Preventive Treatment Alternative for Ileocolic Intussusception With Multiple Recurrences in Children. Surg Laparosc Endosc Percutan Tech. 2018 Oct;28(5):314-317. doi: 10.1097/SLE.0000000000000564. PMID 30067586
- [Background] Yang J, Wang G, Gao J, Zhong X, Gao K, Liu Q, Nan G, Yan C, Chen G, Lu P, Guo C. Liberal surgical laparoscopy reduction for acute intussusception: experience from a tertiary pediatric institute. Sci Rep. 2024 Jan 3;14(1):457. doi: 10.1038/s41598-023-50493-7. PMID 38172223
- [Result] Zhao J, Sun J, Li D, Xu WJ. Laparoscopic versus open reduction of idiopathic intussusception in children: an updated institutional experience. BMC Pediatr. 2022 Jan 17;22(1):44. doi: 10.1186/s12887-022-03112-9. PMID 35038989
- [Result] Li SM, Wu XY, Luo CF, Yu LJ. Laparoscopic approach for managing intussusception in children: Analysis of 65 cases. World J Clin Cases. 2022 Jan 21;10(3):830-839. doi: 10.12998/wjcc.v10.i3.830. PMID 35127899
- [Result] Wei CH, Fu YW, Wang NL, Du YC, Sheu JC. Laparoscopy versus open surgery for idiopathic intussusception in children. Surg Endosc. 2015 Mar;29(3):668-72. doi: 10.1007/s00464-014-3717-1. Epub 2014 Jul 19. PMID 25037726
- [Result] Hill SJ, Koontz CS, Langness SM, Wulkan ML. Laparoscopic versus open reduction of intussusception in children: experience over a decade. J Laparoendosc Adv Surg Tech A. 2013 Feb;23(2):166-9. doi: 10.1089/lap.2012.0174. Epub 2013 Jan 17. PMID 23327343
- [Result] Sklar CM, Chan E, Nasr A. Laparoscopic versus open reduction of intussusception in children: a retrospective review and meta-analysis. J Laparoendosc Adv Surg Tech A. 2014 Jul;24(7):518-22. doi: 10.1089/lap.2013.0415. PMID 24987845
- [Result] Houben CH, Feng XN, Tang SH, Chan EK, Lee KH. What is the role of laparoscopic surgery in intussusception? ANZ J Surg. 2016 Jun;86(6):504-8. doi: 10.1111/ans.13435. Epub 2015 Dec 23. PMID 26699630
- [Result] Benedict LA, Ha D, Sujka J, Sobrino JA, Oyetunji TA, St Peter SD, Fraser JD. The Laparoscopic Versus Open Approach for Reduction of Intussusception in Infants and Children: An Updated Institutional Experience. J Laparoendosc Adv Surg Tech A. 2018 Nov;28(11):1412-1415. doi: 10.1089/lap.2018.0268. Epub 2018 Jul 23. PMID 30036131
- [Result] Takamoto N, Konishi T, Fujiogi M, Kutsukake M, Morita K, Hashimoto Y, Matsui H, Fushimi K, Yasunaga H, Fujishiro J. Outcomes Following Laparoscopic Versus Open Surgery for Pediatric Intussusception: Analysis Using a National Inpatient Database in Japan. J Pediatr Surg. 2023 Nov;58(11):2255-2261. doi: 10.1016/j.jpedsurg.2023.07.004. Epub 2023 Jul 8. PMID 37507337
- [Result] Li N, Bao Q, Yuan J, Zhou X, Feng J, Zhang W. Open transumbilical intussusception reduction in children: A prospective study. J Pediatr Surg. 2021 Mar;56(3):597-600. doi: 10.1016/j.jpedsurg.2020.07.008. Epub 2020 Jul 27. PMID 32792163
- [Result] Jamshidi M, Rahimi B, Gilani N. Laparoscopic and open surgery methods in managing surgical intussusceptions: A randomized clinical trial of postoperative complications. Asian J Endosc Surg. 2022 Jan;15(1):56-62. doi: 10.1111/ases.12965. Epub 2021 Jul 12. PMID 34254449